CLINICAL TRIAL: NCT03081299
Title: Characterization of Bio-psychosocial Pain Profiles in the Perioperative Period
Status: Completed | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 500094-1
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Total Knee Arthroplasty: Descriptive multidimensional tools (the Defense and Veterans Pain Rating Scale (DVPRS) and the electronic Pain Assessment Screening Tool and Outcomes Registry (PASTOR) will be used preoperatively, as an inpatient, and up to 6 months postoperatively.
- Total Hip Arthroplasty: Descriptive multidimensional tools (the Defense and Veterans Pain Rating Scale (DVPRS) and the electronic Pain Assessment Screening Tool and Outcomes Registry (PASTOR) will be used preoperatively, as an inpatient, and up to 6 months postoperatively.
- Mastectomy: Descriptive multidimensional tools (the Defense and Veterans Pain Rating Scale (DVPRS) and the electronic Pain Assessment Screening Tool and Outcomes Registry (PASTOR) will be used preoperatively, as an inpatient, and up to 6 months postoperatively.
- Thoracic Surgery: Descriptive multidimensional tools (the Defense and Veterans Pain Rating Scale (DVPRS) and the electronic Pain Assessment Screening Tool and Outcomes Registry (PASTOR) will be used preoperatively, as an inpatient, and up to 6 months postoperatively.
- Major Abdominal Surgery: Descriptive multidimensional tools (the Defense and Veterans Pain Rating Scale (DVPRS) and the electronic Pain Assessment Screening Tool and Outcomes Registry (PASTOR) will be used preoperatively, as an inpatient, and up to 6 months postoperatively.
- Spinal Fusion: Descriptive multidimensional tools (the Defense and Veterans Pain Rating Scale (DVPRS) and the electronic Pain Assessment Screening Tool and Outcomes Registry (PASTOR) will be used preoperatively, as an inpatient, and up to 6 months postoperatively.

SUMMARY:
This is a prospective descriptive correlational design looking to characterize postoperative pain variables across various procedures that historically have significant levels of persistent post-surgical pain

DETAILED DESCRIPTION:
This is a two institution (Naval Medical Center San Diego and Walter Reed National Military Medical Center) prospective descriptive correlational design looking to characterize postoperative pain variables across various procedures that historically have significant levels of persistent post-surgical pain.

A total goal of 1500 subjects (750 subjects at Walter Reed National Military Medical Center and 750 subjects at Naval Medical Center San Diego) will be queried regarding their postoperative pain experience following mastectomy, thoracic surgery, total knee arthroplasty, total hip arthroplasty, spinal fusion, and major abdominal surgery. Descriptive multidimensional tools (the Defense and Veterans Pain Rating Scale (DVPRS) and the electronic Pain Assessment Screening Tool and Outcomes Registry (PASTOR) will be used preoperatively, as an inpatient, and up to 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 80 and having any of the following surgical procedures: mastectomy, thoracic surgery, total knee arthroplasty, total hip arthroplasty, spinal fusion, and major abdominal surgery.

DEERS eligible

Exclusion Criteria:

* Total Hip/Total Knee arthroplasty revision Younger than 18 years old Refuse participation Cannot understand English Has cognitive deficiencies (subject unable to provide consent for the study, subject unable to complete initial post consent measures)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female military health care beneficiaries age between 18 and 80 years old presenting any of the following surgeries: mastectomy, thoracic surgery, total knee arthroplasty, total hip arthroplasty, spinal fusion, and major abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
DVPRS | perioperatively to 6 months
  To determine how predictive PASTOR/PROMIS measures are for moderate to severe acute postoperative pain as measured by the DVPRS within the first 48 hours postoperatively for all surgical groups and between surgical groups.
PASTOR/PROMIS | perioperatively to 6 months
  To assess any predictive/correlative capability of early postoperative PASTOR/PROMIS measures (7 days,14 days, and 1 month postoperatively) in the prediction of persistent pain at 3 and 6 months for all surgical groups and between surgical groups
Pain phenotypes | perioperatively to 6 months
  To describe various pain phenotypes via multidimensional pain measures throughout the subacute (7 days to 6 months) perioperative period. This description will focus on certain time points but also how such measures change over time (ie pain trajectories)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kent, MD, Principal Investigator — Defense and Veterans Center for Integrative Pain Management
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giordano NA, Kane A, Jannace KC, Rojas W, Lindl MJ, Lujan E, Gelfand H, Kent ML, Highland KB. Discrete and Dynamic Postoperative Pain Catastrophizing Trajectories Across 6 Months: A Prospective Observational Study. Arch Phys Med Rehabil. 2020 Oct;101(10):1754-1762. doi: 10.1016/j.apmr.2020.04.023. Epub 2020 May 21. PMID 32445848